CLINICAL TRIAL: NCT02378194
Title: Change From Baseline to Chronic Kidney Disease Patient Before and After Administration Drug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD-003
Record Dates: First submitted 2015-02-10; First posted 2015-03-04 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2015-02

CONDITIONS: Chronic Renal Failure
Keywords: in stage 3 or 4 steps
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- HD-003 (800mg/day) (Experimental)
  Interventions: Drug: HD-003 (800mg/day)
- HD-003 (1600mg/day) (Experimental)
  Interventions: Drug: HD-003 (1600mg/day)

INTERVENTIONS:
Drug: Placebo — 24 weeks, once daily oral administration
  Arms: Placebo group
Drug: HD-003 (800mg/day) — 24 weeks, once daily oral administration
  Arms: HD-003 (800mg/day)
Drug: HD-003 (1600mg/day) — 24 weeks, once daily oral administration
  Arms: HD-003 (1600mg/day)

SUMMARY:
Chronic renal failure is a syndrome that renal function is decreased, and the patient number is increasing. In addition, patients on dialysis have also increased. Depending on the chronic renal failure aggravated, the deterioration of life caused by the conduct of dialysis patients is caused. In addition, a problem in dialysis treatment is ongoing economic burden surface to increase the life of the patient and family. A solution to this problem is, or stops the progression of chronic renal failure prior to dialysis, it is necessary to delay. As a treatment for inhibiting the progression of chronic renal failure is present, along with diet and blood pressure-lowering drugs or a drug therapy used by kremezin. However, the effect is not enough, new drug development is required.

HD-003 is a novel compound, and found to inhibit the renal failure progression. It was found during the search active substance that appear when the inflammation in animals. The investigators confirmed that the substance is present in the urine of a person during the study, and later established a link between kidney disease hypotheses. When performing the test in animal model renal failure, chronic renal Through the non-clinical testing of the HD-003(general toxicity studies, reproductive, developmental toxicity test, mutagenicity test and antigen tests) showed that a very low toxicity. When going through the review of the safety and pharmacokinetic Phase 1 clinical study, it was confirmed a very satisfactory safety and tolerability. And pharmacokinetic results from the body's absorption in healthy subjects had been done well, a linear correlation was observed. Finally, it was confirmed that the most rapidly excreted into the urine.

This study is a Phase 2a clinical trials performed in patients with chronic renal failure in 3, 4 steps. The evaluation of changes in serum creatinine(sCr) in vivo indicator of renal failure according to the progress. Evaluating the inhibitory effect of HD-003 renal failure progression and dose setting, and to determine the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with chronic renal failure which subjected to conservation therapy.
2. Patient has 15~59mL/min/1.736m2 glomerular filtration rate.
3. Serum creatinine(sCr) is in the range of 1.5~5.0mg/dL at the start of the test and until the start of the test from 52 weeks the serum creatinine is three times more than the number of measurements, and during the final test values of serum creatinine patients with advanced value rises 0.2mg/dL or higher than the first tests.
4. From the start of the test until 52 weeks before the test, serum creatinine the slope of the straight line for the inverse of the value is less than the rare patient -0.0001
5. Inpatient or outpatient
6. Age: 20~75, gender: both

Exclusion Criteria:

1. Patient who start treatment drug or diet that maybe inhibit progress of renal failure within 3 months of the study start
2. Diabetic patients with unstable blood sugar regulation.
3. Patient did not have blood pressure control
4. Patient taking the combination of prohibited substances
5. Dialysis patient
6. Patient with gout
7. Patient who merged with a progressive muscular dystrophy, polymyositis, etc.
8. Patients with symptoms of cerebral vascular disorders
9. Women who are pregnant or breast-feeding
10. Patient with infectious disease
11. Patient with gastric ulcer
12. Patients who has difficult diet, medication, etc.
13. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
14. Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
serum creatinine rate inverse number's change | up to 24 weeks
GFR measurements (confirmed by the method MDRD via the value of sCr) | up to 24 weeks

OTHER OUTCOMES:
Number of Participants with Adverse Events | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Choi, Principal Investigator — Yonsei University Health System, Severance Hospital